CLINICAL TRIAL: NCT07377812
Title: Predictors of Length of Stay and Days Alive and at Home Within 30 Days (DAH30) After Elective Minimally Invasive Surgery in Older Adults: A Multicenter Retrospective Observational Study With International External Validation
Brief Title: Predictors of Length of Stay and DAH30 After Elective Minimally Invasive Surgery in Older Adults
Acronym: HOME-30
Status: Completed | Type: Observational
Sponsor: Dmitrii Semenov (Other)
Responsible Party: Sponsor-Investigator, Dmitrii Semenov, Consultant Surgeon, Dmitrii Semenov
Other Study IDs: HOME30-RETRO
Record Dates: First submitted 2026-01-20; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Recovery
Keywords: Older adults; Minimally invasive surgery; Days alive and at home; Postoperative recovery
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older Adults Undergoing Elective Minimally Invasive Surgery: This cohort includes adults aged 70 years and older who underwent elective minimally invasive surgical procedures. The study is retrospective and observational in nature. No interventions were assigned as part of the study; all analyses are based on routinely collected clinical data obtained during standard care.
  Interventions: Other: No Intervention (Observational Study)

INTERVENTIONS:
Other: No Intervention (Observational Study) — This is a retrospective observational study. No interventions were assigned or administered as part of the study. All analyses are based on routinely collected clinical data obtained during standard clinical care.

SUMMARY:
This retrospective observational study aims to evaluate short-term postoperative outcomes in older adults undergoing elective minimally invasive surgery. The primary focus is on patient-centered recovery measures, including length of hospital stay and the number of days patients are alive and at home within 30 days after surgery.

Using routinely collected clinical data, the study will assess demographic, clinical, and perioperative factors associated with delayed discharge and reduced time spent at home after surgery. Understanding these factors may help clinicians and healthcare systems better plan postoperative care and optimize recovery pathways for older surgical patients.

DETAILED DESCRIPTION:
This is a multicenter, retrospective, observational cohort study designed to identify predictors of short-term postoperative outcomes in older adults undergoing elective minimally invasive surgical procedures.

The study includes patients aged 70 years and older who underwent elective laparoscopic or minimally invasive abdominal surgery. All data are derived exclusively from routinely collected medical records generated during standard clinical care. No study-related interventions, changes in clinical management, or additional patient contacts are performed.

The primary outcomes of interest are length of hospital stay and days alive and at home within 30 days after surgery (HOME-30 / DAH30). Secondary analyses explore the association of demographic characteristics, comorbidities, perioperative factors, and discharge timing with these outcomes.

The study aims to improve understanding of non-medical contributors to prolonged hospitalization in older surgical patients and to support the development of patient-centered outcome measures applicable across different healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 years or older at the time of surgery
* Undergoing elective minimally invasive surgical procedures
* Surgery performed under general anesthesia
* Availability of complete medical records required to assess study outcomes

Exclusion Criteria:

* Emergency or urgent surgical procedures
* Open (non-minimally invasive) surgery
* Incomplete medical records precluding outcome assessment

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adult patients aged 70 years and older who underwent elective minimally invasive surgical procedures under general anesthesia in participating centers. All data are collected retrospectively from routine clinical records.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-01 (Actual); Study Completion 2026-01 (Actual)

PRIMARY OUTCOMES:
Days Alive and at Home Within 30 Days After Surgery (DAH30) | Postoperative Day 0 through Postoperative Day 30
  Days Alive and at Home within 30 days after surgery (DAH30), defined as the total number of days during the first 30 days following the index surgical procedure that the patient is alive and not admitted to an acute care hospital.

SECONDARY OUTCOMES:
Length of Hospital Stay After Surgery | Perioperative period
  Length of hospital stay, defined as the number of days from the date of surgery to the date of discharge from the index hospitalization.
All-Cause Hospital Readmission Within 30 Days After Surgery | Postoperative Day 1 through Postoperative Day 30
  Any unplanned hospital readmission for any cause occurring within 30 days after discharge from the index surgical hospitalization.
Postoperative Complications Within 30 Days | Postoperative Day 0 through Postoperative Day 30
  Occurrence of postoperative complications within 30 days after surgery, classified according to the Clavien-Dindo grading system.
Discharge Destination After Surgery | Perioperative period
  Discharge destination following index hospitalization, categorized as home, rehabilitation facility, skilled nursing facility, or other healthcare institution.

CONTACTS AND LOCATIONS:
Locations (1):
- K+31 Clinic, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in the published articles, including demographic characteristics, perioperative variables, comorbidities, surgical details, and outcome measures such as DAH30, length of hospital stay, postoperative complications, readmissions, and discharge destination.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 6 months after publication, with no end date.
Access Criteria: Data will be shared upon reasonable request. Requests should include a brief research proposal and will be reviewed by the study investigators. Data will be provided for non-commercial academic research purposes only, following approval and execution of a data use agreement. All shared data will be fully de-identified.